CLINICAL TRIAL: NCT05671770
Title: Study Based on Electronic Health RecOrds to Identify Patients at High-risk of Fabry DiseasE
Brief Title: Study Based on Electronic Health RecOrds to Identify Patients at High-risk of Fabry DiseasE (HOPE Fabry)
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17546
Record Dates: First submitted 2022-12-20; First posted 2023-01-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Patients with chronic kidney disease
- Cohort 2: Patients with hypertrophic cardiomyopathy

SUMMARY:
Primary objective:

To estimate the prevalence of patients who are at high-risk for Fabry Disease (FD) in the Cleveland Clinic, Abu Dhabi (CCAD) United Arab Emirates (EMR) database from May 2016 to May 2022, according to the predictive algorithm (i.e., feasibility assessment eligibility criteria)

Secondary objectives:

* To estimate the prevalence of FD among patients at high-risk for FD (i.e., among enrolled patients)
* To characterize the patient profile, overall and in Cohorts 1 and 2
* To describe the most common characteristics among positive FD patients and negative FD patients

DETAILED DESCRIPTION:
Patients at high-risk for FD will be consecutively enrolled over approximately 6 months

ELIGIBILITY:
Inclusion Criteria:

* Patients who were identified as high-risk for FD via the predictive algorithm per the feasibility assessment
* Patients who have signed an informed consent form

Cohort 1 (chronic kidney disease)

* Adult male patient ≤60 years old or adult female patient of any age
* Having chronic kidney disease
* Having proteinuria
* Having one or more of the following conditions:

  * Neuralgia and neuritis, unspecified
  * Disturbances in skin sensation
  * Anhidrosis, and
  * Hypertrophic cardiomyopathy.

Cohort 2 (hypertrophic cardiomyopathy)

* Adult male patient ≤50 years old or adult female patient of any age
* Having hypertrophic cardiomyopathy
* Having one or more of the following conditions:

  * transient cerebral ischemic attack,
  * chronic kidney disease.

Exclusion Criteria:

* Patients with an established diagnosis of FD.
* Pregnant subject at the time of the study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease (Cohort 1) or hypertrophic cardiomyopathy (Cohort 2), who fulfill the criteria for being at high-risk for FD, per the predictive algorithm, and provide informed consent, will be eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Number and proportion of patients at high-risk for FD in the CCAD EMR database | Up to 6 months
  The prevalence of patients at high-risk for FD in the CCAD EMR database, according to the predictive algorithm, from May 2016 to May 2022, will be estimated. The percentage (and 95% confidence interval [CI]) of patients at high-risk for FD will be calculated, overall and in Cohorts 1 and 2.

SECONDARY OUTCOMES:
Number and proportion of patients with FD (overall and among patients in Cohorts 1 and 2) | Up to 6 months
  The prevalence of patients diagnosed with FD among patients at high-risk for FD (i.e., among enrolled patients) will be estimated. The percentage (and 95% CI) of patients diagnosed with FD will be calculated, overall and in Cohorts 1 and 2.
To describe the following patient characteristics, overall and in Cohorts 1 and 2: | Up to 6 months
  The following patient characteristics will be summarized by descriptive statistics, overall and in Cohorts 1 and 2: demographics, physical examinations, medical history, comorbidities, concomitant medications, clinical symptoms, and FD diagnostic test results including test outcome for FD (positive/negative).
To describe the following patient characteristics, among positive FD patients and negative FD cases: | Up to 6 months
  The following patient characteristics will be summarized by descriptive statistics, among positive FD patients and negative FD patients: demographics, physical examinations, medical history, comorbidities, concomitant medications, and clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Cleveland Clinic AbuDhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org